CLINICAL TRIAL: NCT02725528
Title: A Multi-Center, Randomized Controlled Trial Comparing The Clinical Effectiveness and Cost-Effectiveness of Collagenase Injection (Xiaflex) and Palmar Fasciectomy in the Management of Dupuytren's Disease
Brief Title: Evaluation of Xiaflex: Trial of Effectivenss iN Dupuytren's
Acronym: EXTEND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Principal Investigator, Achilleas Thoma, Dr. Achllieas Thoma, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSI 2016-03
Record Dates: First submitted 2016-03-22; First posted 2016-04-01 (Estimated); Results first posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-06

CONDITIONS: Dupuytren's Disease
MeSH Terms: conditions — Dupuytren Contracture | interventions — Collagenases; Enzymes; Microbial Collagenase

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- collagenase injection (Active Comparator): This procedure will be performed either in a minor procedure room or the hand clinic as per surgeon's routine practice. Collagenase will be administered with or without local anesthesia. As this is a pragmatic study there may be more than one digit injected at a time just as surgery occurs on more than one digit at a time. A recently published study by Gaston et al confirmed that two concurrent injections of collagenase to 2 affected joints in the same hand are generally well tolerated and the frequency of most adverse events (AEs) is similar to those reported in studies that use single sequential injections.
  Interventions: Drug: collagenase injection
- limited palmar fasciectomy (Active Comparator): The Dupuytren's cord will be excised under local anesthesia in a minor procedure room setting or main operating room under local or general anesthetic depending on the complexity of the disease and the surgeon's routine. As this is a pragmatic study comparison of collagenase injections (novel intervention) to limited palmar fasciectomy as it is actually presently performed in all settings academic or community (local in minor room or general/local anesthetic in the main operating room) will be examined. Surgery will be performed according to the operating surgeon's preferred technique i.e. zig-zag Brunner incision or straight incision with z-plasty closure of the skin.
  Interventions: Procedure: limited palmar fasciectomy

INTERVENTIONS:
Drug: collagenase injection — injection
  Other Names: enzyme, collagenase clostridium histolyticum, xiaflex
  Arms: collagenase injection
Procedure: limited palmar fasciectomy — surgery
  Arms: limited palmar fasciectomy

SUMMARY:
This is a prospective, multi-centre, pragmatic randomized controlled trial to compare both the clinical effectiveness and cost-effectiveness of collagenase injections (CI) versus limited palmar fasciectomy (LPF) to determine if collagenase is a superior treatment in terms of improved quality of life and reducing recurrence of the disease without serious complications. Since collagenase injections are costly it is also important to know if this novel intervention is cost-effective from the patient, Ministry of Health and societal perspectives.

DETAILED DESCRIPTION:
Limited palmar fasciectomy (LPF) and collagenase injection (CI) are the most common procedures to manage symptoms of Dupuytren's Disease. This randomized controlled trial (RCT) aimed to directly compare patient outcomes 12 months following CI and LPF. Twenty-two patients with Dupuytren's Disease were randomized to either LPF or CI. The primary outcome was health state measured by the Michigan Hand Questionnaire. Secondary outcomes were health status (The Health Utility Index-3), function (The Unité Rhumatologique des Affections de la Main and The Southampton Dupuytren's Scoring Scheme), and range of motion (ROM) of treated digits. Measurements were collected at baseline and 1-, 3-, 6-, and 12-months post-procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Canadian Citizen
2. 18 years of age or older
3. Dupuytren's contracture of the metacarpophalangeal (MCP) joint or of the proximal interphalangeal (PIP) joint with a fixed flexion contracture of 20º or greater in at least 1 finger (not the thumb)
4. Demonstrated inability to simultaneously place the affected finger and palm flat on a table
5. Able to understand and communicate in English

Exclusion Criteria:

1. Previous treatment of the primary joint within 90 days of study inclusion
2. Patients undergoing any concomitant procedure on the same hand (e.g. carpal tunnel release, stenosing tenosynovitis release)
3. Persistent extension deficit from a previous surgery of the same digit
4. Any chronic muscular or neuromuscular disorder affecting wrist or hand
5. Patient generally unfit for surgery
6. Patient with specific treatment preference
7. Bleeding disorder or recent stroke
8. Allergy to collagenase
9. Collagenase treatment or treatment with any investigational drug within 30 days of study inclusion
10. Use of a tetracycline derivative within 14 days of first dose of study drug (because tetracycline derivatives may inhibit the collagenolytic activity of mammalian collagenase homologs [i.e., matrix metalloproteinases])
11. Pregnant or breast feeding patients
12. Patients who do not have insurance coverage for collagenase injections
13. Patients who are unable to provide informed consent or are unable to complete quality of life questionnaires due to mental capacity or neuro-psychological problems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-07-08 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Achilleas Thoma, MD MSc FRCSC, Principal Investigator — McMaster University
Locations (10):
- Canada (10):
  - Hamilton Health Sciences, Hamilton, Ontario
  - St. Joseph's Healthcare / McMaster University, Hamilton, Ontario
  - St. Joseph's Hospital, Hamilton, Ontario
  - St. Joseph's Healthcare, London, Ontario
  - Markham Stouffville Hospital, Markham, Ontario
  - 679 Davis St. Suite 209, Newmarket, Ontario
  - Halton Healthcare Services, Oakville, Ontario
  - Oakville Trafalgar Hospital, Oakville, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - North York General Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Collagenase Injection: This procedure was performed either in a minor procedure room or the hand clinic as per surgeon's routine practice. Collagenase will be administered with or without local anesthesia. As this was a pragmatic study, if injection was required in more than one digit, this was done, as per standard of care.
  The patient's affected hand was prepped with antiseptic solution. Using a hubless syringe with 0.01 mL graduations and a permanently fixed 26- or 27-gauge ½ inch needle the required amount of reconstituted collagenase clostridium histolyticum was withdrawn as follows:
  1. Cord affecting an MP joint, withdraw 0.25 mL of the reconstituted solution;
  2. Cord affecting a PIP joint: withdraw 0.20 mL of the reconstituted solution per published guidelines.
  collagenase injection: injection
- Limited Palmar Fasciectomy: The Dupuytren's cord was excised in a minor procedure room setting or main operating room under local or general anesthetic depending on the complexity of the disease and the surgeon's routine. The procedure was performed according to the surgeon's preferred technique (i.e., zig-zag Brunner incision or straight incision with z-plasty closure of the skin). Loupe magnification was used in surgery to identify and protect the digital neurovascular bundles. The diseased Dupuytren's fascia (cords) causing the contracture was excised. Contracted ligaments at the PIP joints were released by passive stretching or with knife intraoperatively. A plaster splint was applied at the discretion of the surgeon.
  limited palmar fasciectomy: surgery
Period: Overall Study
Arm/Group | Collagenase Injection | Limited Palmar Fasciectomy
Started | 8 (Number of participant's randomized to this group.) | 14 (Number of participant's randomized to this group.)
Completed | 7 (Completed primary outcome at 12 months (i.e., Michigan Hand Questionnaire).) | 9 (Completed primary outcome at 12 months (i.e., Michigan Hand Questionnaire).)
Not Completed | 1 | 5
Not completed — Lost to Follow-up | 1 | 4
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: One participant in the limited palmar fasciectomy (LPF) group dropped out immediately after randomization, before baseline outcomes were measured, thus the size of the LPF group is 13, not 14.
Groups:
- Total: Total of all reporting groups
Arm/Group | Collagenase Injection | Limited Palmar Fasciectomy | Total
Number analyzed (Participants) | 8 | 13 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (10.2) | 65 (9) | 65.3 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 7 | 11 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 8 | 13 | 21
Affected Hand [Count of Participants; unit: Participants]
  Right | 6 | 9 | 15
  Left | 2 | 4 | 6
Affected Digit [Count of Participants; unit: Participants]
  Little | 2 | 8 | 10
  Ring | 1 | 3 | 4
  Long | 1 | 0 | 1
  Little & Ring | 4 | 0 | 4
  Long & Little | 0 | 1 | 1
  Little, Ring & Long | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Health-related Quality of Life (HRQL) Using the Michigan Hand Outcomes Questionnaire (MHQ)
Description: Michigan Hand Outcomes Questionnaire (MHQ). Converted to a score rated 0-100 (where higher scores represent better function).
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Collagenase Injection | Limited Palmar Fasciectomy
Number analyzed (Participants) | 7 | 9
units on a scale | 78.1 (14.9) | 68.3 (15.7)
Statistical Analysis 1: Comparison: Collagenase Injection vs Limited Palmar Fasciectomy; Between groups analysis for PROMs, QALYs and ROM at 12-months were determined using one-way analysis of covariance (ANCOVA). Group was entered as the independent variable, the 12-month outcome of interest was entered as the dependent variable and the baseline value for the corresponding outcome measure was entered as the covariate. Statistical significance was considered at p < .05; all analyses were performed using SPSS® version 26.0; Test type: Superiority; p = 0.05, ANCOVA

2. Secondary Outcome: HRQL Measured With the Health Utility Index Mark 3 (HUI3) of Health
Description: Health Utility Index Mark 3 (HUI3) of Health. The HUI3 is a generic multi-attribute health-status classification instrument composed of eight attributes or dimensions: vision, hearing, speech, ambulation, dexterity, emotion, cognition, and pain with five or six levels per attribute. Dimensions are combined to produce one health utility score. The HUI3 produces health utilities anchored at 0 (minimum) for equal to being dead and 1 (maximum) for perfect health.
Time Frame: 1 year
Population: Missing data addressed by using available case analysis. Difference from flow chart due to participant's loss to follow up. Number of participant's in limited palmar fasciectomy group includes 1 additional participant who completed this outcome, but did not complete the primary outcome as indicated in the participant flow chart.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Collagenase Injection | Limited Palmar Fasciectomy
Number analyzed (Participants) | 7 | 10
units on a scale | 0.8 (0.79) | 0.79 (0.14)
Statistical Analysis 1: Comparison: Collagenase Injection vs Limited Palmar Fasciectomy; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.05, ANCOVA

3. Secondary Outcome: HRQL Measured With the Unité Rhumatologique Des Affections de la Main (URAM)
Description: Unité Rhumatologique des Affections de la Main (URAM). The URAM is a disease-specific HRQL measure developed for Dupuytren's Disease (DD) and is composed of a 9-item patient-reported questionnaire. Each item is scored between 0 and 5 depending on the difficulty in performing that particular function with total scores for DD-associated disability ranging from 0 (best) to 45 (worst). High scores suggest high levels of disability and disturbance. The URAM scale is a 1-domain outcome measure postulated to be related to disability associated with DD.
Time Frame: 1 year
Population: Missing data addressed by using available case analysis. Difference from flow chart due to incomplete data collection for this outcome (i.e. loss to follow up).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Collagenase Injection | Limited Palmar Fasciectomy
Number analyzed (Participants) | 5 | 9
units on a scale | 4.6 (9.2) | 5.2 (7.6)
Statistical Analysis 1: Comparison: Collagenase Injection vs Limited Palmar Fasciectomy; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.05, ANCOVA

4. Secondary Outcome: HRQL Measured With the Southampton Dupuytren's Scoring Scheme (SDSS)
Description: The SDSS is disease-specific scoring system developed for Dupuytren's Disease (DD) with 5 domains, each relevant to DD and scored on a five-point scale (no problem, mild inconvenience, modest inconvenience, definitely troublesome, severe problem). The minimum score is 0 and maximum score is 20 with higher scores suggesting higher levels of disability.
Time Frame: 1 year
Population: Missing data addressed by using available case analysis. Difference from flow chart due to incomplete data collection for this outcome (i.e. loss to follow up). Number of participant's in limited palmar fasciectomy group includes 1 additional participant who completed this outcome, but did not complete the primary outcome as indicated in the participant flow chart.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Collagenase Injection | Limited Palmar Fasciectomy
Number analyzed (Participants) | 6 | 10
units on a scale | 6.5 (3.2) | 7.2 (3.7)
Statistical Analysis 1: Comparison: Collagenase Injection vs Limited Palmar Fasciectomy; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.05, ANCOVA

5. Secondary Outcome: Quality Adjusted Life Years (QALY) Measured With the Health Utility Index Mark 3 (HUI3)
Description: QALY was calculated by multiplying the difference between quality of life, as measured by the HUI-3 score before and after the intervention by the remaining years of life of the average patient (i.e., life expectancy - patient's age). Life expectancy was set at 79 years for males, and 84 years for females. Higher QALYs represent improved (better) patient outcomes.
Time Frame: 1 year
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: quality-adjusted life years
Arm/Group | Collagenase Injection | Limited Palmar Fasciectomy
Number analyzed (Participants) | 7 | 10
quality-adjusted life years | 0.83 (1.7) | 0.93 (2.8)
Statistical Analysis 1: Comparison: Collagenase Injection vs Limited Palmar Fasciectomy; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.05, ANCOVA

6. Secondary Outcome: Recurrence Rates
Description: Reccurence was measured as whether or not participants received a repeat diagnosis of Dupuytren's disease with loss of finger extension at the site of prior intervention and underwent palmar fasciectomy (following the collagenase injection or as a revision operation) after initial study treatment. The time horizon for recurrence was between 1-4 years post initial study treatment. Outcome was dichotomous (i.e., recurrence; yes or no).
Time Frame: 1-4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Collagenase Injection | Limited Palmar Fasciectomy
Number analyzed (Participants) | 7 | 9
Participants | 3 | 1
Statistical Analysis 1: Comparison: Collagenase Injection vs Limited Palmar Fasciectomy; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.05, ANCOVA

7. Secondary Outcome: Loss of Extension MCP
Description: Passive range of motion degree of extension was measured using a goniometer. Difference in degree, as measured by a goniometer, between the participant's resting maximum extension of the metacarpal-phalangeal joint, relative to a metacarpal-phalangeal joint at full extension (i.e., 0 degrees)
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Collagenase Injection | Limited Palmar Fasciectomy
Number analyzed (Participants) | 7 | 9
Degrees | 20 (26.9) | 2.56 (3.97)
Statistical Analysis 1: Comparison: Collagenase Injection vs Limited Palmar Fasciectomy; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.05, ANCOVA

8. Secondary Outcome: Loss of Extension PIP
Description: Passive range of motion degree of extension was measured using a goniometer. Difference in degree, as measured by a goniometer, between the participant's resting maximum extension of the proximal inter-phalangeal joint, relative to a proximal inter-phalangeal joint at full extension (i.e., 0 degrees)
Time Frame: 1 year
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Collagenase Injection | Limited Palmar Fasciectomy
Number analyzed (Participants) | 5 | 9
Degrees | 23.2 (18.17) | 17.2 (21.81)
Statistical Analysis 1: Comparison: Collagenase Injection vs Limited Palmar Fasciectomy; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.05, ANCOVA

9. Secondary Outcome: Loss of Extension DIP
Description: Passive range of motion degree of extension was measured using a goniometer. Difference in degree, as measured by a goniometer, between the participant's resting maximum extension of the distal inter-phalangeal joint, relative to a distal inter-phalangeal joint at full extension (i.e., 0 degrees)
Time Frame: 1 year
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Collagenase Injection | Limited Palmar Fasciectomy
Number analyzed (Participants) | 1 | 2
Degrees | 8 (0) | 10 (14.14)
Statistical Analysis 1: Comparison: Collagenase Injection vs Limited Palmar Fasciectomy; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.05, ANCOVA

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Collagenase Injection | Limited Palmar Fasciectomy
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/13
Other Adverse Events (participants affected / at risk) | 0/8 | 0/13

LIMITATIONS AND CAVEATS:
Limitations include small sample size, poor recruitment (due health insurance coverage, treatment preference, and the discontinuation of Xiaflex® in Canada), and poor response rate and outcome data collection due to onset and restriction associated with COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-07): https://cdn.clinicaltrials.gov/large-docs/28/NCT02725528/Prot_SAP_000.pdf